CLINICAL TRIAL: NCT01532778
Title: Perception Ortho-nasale du Gras Chez l'Homme Sain : Relations Entre Typages olfactométriques, Sensoriels et Composition de la Salive.
Brief Title: Saliva Modification Related to Fat Perception in Human
Acronym: SensInFat
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A01225-34
Record Dates: First submitted 2012-02-10; First posted 2012-02-14 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Fat Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The perception of fat represents major scientific and nutritional issues. This research aims to identify salivary markers that could predict and possibly explain this perception in healthy human being. This would help to develop nutritional strategies for a more rational consumption of fat.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-60 years

Exclusion Criteria:

* Female
* Non healthy

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male, healthy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CSGA, Dijon, France

IPD SHARING:
Plan to Share IPD: No